CLINICAL TRIAL: NCT04778150
Title: Relationship Between Non-Invasive Measurement of Jugular Venous Oxygen Saturation (SjvO2) Using Near Infraread Spectroscopy and Measurement of Mixed Venous Saturation of Oxygen (SvO2) in Patients Undergoing Liver Transplantation Surgery
Brief Title: Non-Invasive Measurement of SjvO2 Using Near Infrared Spectroscopy in Patients Undergoing Liver Transplantation Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Eduardo Schiffer, MD, PhD, University Hospital, Geneva
Other Study IDs: SJVO2 vs SVO2
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2022-05

CONDITIONS: Impaired Oxygen Delivery; Transplant; Failure, Liver
Keywords: SvO2; SjvO2; Portal vein clamping; Liver transplantation surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: VO 100 medical device from Mespere LifeSciences — The investigators want to show a positive relationship between SjvO2 and SvO2 in order to possibly use in the future SjvO2 measured by VO 100 as a noninvasive surrogate of SvO2 in patients undergoing liver transplantation surgery.

SUMMARY:
Mixed venous oxygen saturation (SvO2) is an important parameter in the management of patient during liver transplantation surgery especially during portal vein clamping. The only way to measure it is to use a pulmonary artery catheter. If the authors can show a positive relationship between invasive SvO2 measurement and noninvasive jugular venous oxygen saturation (SjvO2) measurement with VO 100 medical device, it will possible to use SjvO2 as a noninvasive surrogate of SvO2 in patients during liver transplantation surgery.

DETAILED DESCRIPTION:
SvO2 measures mixed venous oxygen saturation from the lower and upper half of the body. To be measured, Sv02 requires a central venous catheter. SvO2 gives knowledge about the balance between the delivery of oxygen and oxygen consumption in the body. Interest in SvO2 monitoring in anesthesia and critical care has been debated. However, SvO2 is still recommended as a major hemodynamic target of early resuscitation of critically ill patients. SvO2 measurement through pulmonary artery catheter is accompanied with morbidity due to its invasiveness. During liver transplantation surgery, measurement of SvO2 is required to adequately manage hemodynamics of the patient, especially during portal venous clamping.

VO 100 medical device from Mespere LifeSciences allows a non-invasive measurement of SjvO2 using the NIRS technique. Jugular venous oxygen saturation (SjvO2) is a measurement of the amount of oxygen left in the venous system after the brain has removed the oxygen that it needs.

On the same principle that a positive relationship between ScvO2 and SvO2 has been shown, what the investigators are trying to do is to show a positive relationship between SjvO2 and SvO2 in order to possibly use in the future SjvO2 measured by VO 100 as a noninvasive surrogate of SvO2 during liver transplantation surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients routinely equipped with a pulmonary artery catheter just before liver transplantation surgery allowing SvO2 measurement.

Exclusion Criteria:

* Adult patients not equipped with pulmonary artery catheter for liver transplantation surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing liver transplantation surgery for whom measurement of SvO2 is required especially during portal vein clamping.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Comparison of venous oxygen saturation | Continuously during liver transplantation surgery
  Comparison of SvO2 values from pulmonary artery catheter blood and SjvO2 values from the VO 100 (% oxygen saturation)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Schiffer, MD, Principal Investigator — Head of anesthesia for liver transplantation surgery
Locations (1):
- University of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No